CLINICAL TRIAL: NCT02903914
Title: Safety, Pharmacokinetics, and Pharmacodynamics of Escalating Oral Doses of the Arginase Inhibitor INCB001158 (Formerly Known as CB1158) as a Single Agent and in Combination With Immune Checkpoint Therapy in Patients With Advanced/Metastatic Solid Tumors
Brief Title: Arginase Inhibitor INCB001158 as a Single Agent and in Combination With Immune Checkpoint Therapy in Patients With Advanced/Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: INCB 01158-101; Mk3475 Keynote 741 (Other: Merck); 2017-002903-82 (EudraCT Number)
Record Dates: First submitted 2016-09-09; First posted 2016-09-16 (Estimated); Results first posted 2021-09-30 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Cancer; Solid Tumors; Colorectal Cancer (CRC); Gastric Cancer; Head and Neck Cancer; Lung Cancer; Renal Cell Carcinoma (RCC); Bladder Cancer; UC (Urothelial Cancer); Mesothelioma
Keywords: Immuno-Oncology; Checkpoint Inhibitors; Tumor Metabolism; Programmed cell death protein-1 (PD-1) inhibitor; Programmed death ligand 1 (PD-L1) inhibitor; Solid Tumors; RCC; MEL; NSCLC; Arginase; Arginase Inhibitor; INCB001158 (CB-1158); SCCHN; GEJ; Immune Therapy
MeSH Terms: conditions — Neoplasm Metastasis; Colorectal Neoplasms; Stomach Neoplasms; Head and Neck Neoplasms; Lung Neoplasms; Carcinoma, Renal Cell; Urinary Bladder Neoplasms; Mesothelioma; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — CB-1158; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- INCB00158 was administered as monotherapy at 50mg twice daily (Experimental): Monotherapy Part 1a: INCB001158 administered orally in patients with advanced/metastatic solid tumors. Escalating doses will be explored to determine the recommended phase 2 dose (RP2D).
  Interventions: Drug: INCB001158
- INCB00158 was administered as monotherapy at 75mg twice daily (Experimental): Monotherapy Part 2a: INCB001158 administered orally at the RP2D in patients with advanced/metastatic NSCLC (EGFR and Anaplastic Lymphoma Kinase (ALK) negative) previously treated with Standard of Care (SOC).
  Interventions: Drug: INCB001158
- INCB00158 was administered as monotherapy at 100mg twice daily (Experimental): Monotherapy Part 2b: INCB001158 administered orally at the RP2D in patients with advanced/metastatic CRC previously treated with SOC.
  Interventions: Drug: INCB001158
- INCB00158 was administered as monotherapy at 150mg twice daily (Experimental): Monotherapy Part 2c: INCB001158 administered orally at the RP2D in patients with Bladder Cancer, Gastric or Gastroesophageal Junction (GEJ) Cancer, Renal Cell Cancer (RCC), Squamous Cell Carcinoma of the Head and Neck (SCCHN), Urothelial Cell Cancer (UCC), or Melanoma, previously treated with SOC.
  Interventions: Drug: INCB001158
- INCB00158 was administered in combination with pembroluzimab at 50mg twice daily (Experimental): Monotherapy Part 2d: INCB001158 administered orally at the RP2D in patients with any tumor types in Parts 2a, 2b, or 2c.
  Interventions: Drug: INCB001158
- INCB00158 was administered in combination with pembroluzimab at 75mg twice daily (Experimental): Combination Part 1b: INCB001158 and Pembrolizumab administered in patients with advanced/metastatic NSCLC, Melanoma, Urothelial Cell Cancer, MSI CRC, MSS CRC, Gastric or Gastroesophageal Junction (GEJ) Cancer, SCCHN and Mesothelioma. Multiple dose levels will be explored to determine the recommended phase 2 dose (RP2D).
  Interventions: Drug: INCB001158; Drug: Pembrolizumab
- INCB00158 was administered in combination with pembroluzimab at 100mg twice daily (Experimental): Part 3a: INCB001158 and Pembrolizumab the combination RP2D in patients with advanced/metastatic NSCLC (EGFR and ALK negative) with disease progression on anti-PD-1 therapy or prolonged stable disease on Pembrolizumab in the immediate prior line of therapy.
  Interventions: Drug: INCB001158; Drug: Pembrolizumab
- INCB001158 50 mg BID in combination with pembrolizumab (Experimental): Part C: evaluated a reduced dose of INCB001158 50 mg BID in combination with pembrolizumab with patients with moderately impaired renal function.
  Interventions: Drug: INCB001158; Drug: Pembrolizumab

INTERVENTIONS:
Drug: INCB001158 — Arginase Inhibitor
  Other Names: CB-1158
Drug: Pembrolizumab — PD-1 Inhibitor
  Other Names: Keytruda
  Arms: INCB001158 50 mg BID in combination with pembrolizumab; INCB00158 was administered in combination with pembroluzimab at 100mg twice daily; INCB00158 was administered in combination with pembroluzimab at 75mg twice daily

SUMMARY:
This study is an open-label Phase 1/Phase 2 evaluation of INCB001158 as a single agent and in combination with immune checkpoint therapy in patients with advanced/metastatic solid tumors.

DETAILED DESCRIPTION:
This study is an open-label Phase 1 evaluation of INCB001158 as a single agent and in combination with immune checkpoint therapy in patients with advanced/metastatic solid tumors.

Single Agent INCB001158:

Patients with advanced/metastatic solid tumors will be enrolled into escalating monotherapy dose cohorts to determine the Recommended Phase 2 Dose (RP2D) of INCB001158. Additional patients with NSCLC, Colorectal Cancer (CRC), and other tumors including SCCHN, RCC, Gastric, Bladder and Melanoma will be enrolled at the single agent RP2D.

Combination Treatment:

Patients with advanced/metastatic NSCLC, Melanoma, Urothelial, Microsatellite Instability (MSI)/ Microsatellite Stable (MSS) CRC, Gastric, SCCHN and Mesothelioma will be enrolled into separate cohorts of combination therapy (INCB001158 and Pembrolizumab) to determine the RP2D.

In the dose expansion phase, additional patients with NSCLC, Melanoma, Urothelial, MSI/MSS CRC, Gastric, SCCHN and Mesothelioma will be treated with the combination of INCB001158 and Pembrolizumab at the RP2D.

All patients will be assessed for safety, pharmacokinetics, biomarkers and tumor response.

ELIGIBILITY:
*Additional cohort specific criteria may apply

Inclusion Criteria:

* Must be age 18 or older
* Ability to provide written informed consent in accordance with federal, local, and institutional guidelines
* Histological or cytological diagnosis of metastatic cancer or locally advanced cancer that is not amenable to local therapy
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
* Life Expectancy of at least 3 months
* Adequate hepatic, renal (moderately impaired renal function in cohort 1c only), cardiac, and hematologic function
* Measurable disease by RECISTv1.1 criteria
* Resolution of treatment-related toxicities
* Willingness to avoid pregnancy or fathering children
* Prior anti-PD-1 treatment for combination dose expansion cohorts 1c, 3a - 3d

Exclusion Criteria:

* Currently pregnant or lactating
* Unable to receive oral medications
* Unable to receive oral or IV hydration
* Intolerance to prior anti-PD-1/PD-L1 therapy
* Prior anti-PD-1 treatment for combination dose expansion cohorts 1c, 3e - 3h
* Prior severe hypersensitivity reaction to another monoclonal antibody (mAb)
* Any other current or previous malignancy within 3 years except protocol allowed malignancies
* Chemotherapy, Tyrosine Kinase Inhibitor therapy, radiation therapy or hormonal therapy within 2 weeks
* Immunotherapy or biological therapy, or investigational agent within 3 weeks (Note: some cohort exceptions allow anti-PD-1 therapy)
* Active known or suspected exclusionary autoimmune disease
* Any condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other systemic immunosuppressive medications within 2 weeks
* Concomitant therapy with valproic acid/valproate-containing therapies
* Concomitant therapy with allopurinol and other xanthine oxidase inhibitors
* History of known risks factors for bowel perforation
* Symptomatic ascites or pleural effusion
* Major surgery within 28 days before Cycle 1 Day 1
* Active infection requiring within 2 weeks prior to first dose of study drug
* Patients who have HIV, Hepatitis B or C
* Conditions that could interfere with treatment or protocol-related procedures
* Active, non-stable brain metastases or CNS disease
* Known deficiencies or suspected defect in the urea cycle
* Received live-virus vaccination within 30 days (seasonal flu vaccine allowed if non-live virus)
* NSCLC with EGFR or ALK mutation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2016-09-14 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2022-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emil Kuriakose, MD, Study Director — Calithera Biosciences, Inc; Sven Gogov, MD, Study Director — Incyte Corporation
Locations (19):
- United States (12):
  - University of South Alabama, Mobile, Alabama
  - Honor Health/Pinnacle Oncology Hematology, Scottsdale, Arizona
  - University of Arizona, Tucson, Arizona
  - Georgetown, Washington D.C., District of Columbia
  - Johns Hopkins, Baltimore, Maryland
  - BIDMC, Boston, Massachusetts
  - DFCI, Boston, Massachusetts
  - Henry Ford, Detroit, Michigan
  - Sarah Cannon Research Institute at Tennessee Oncology, Nashville, Tennessee
  - Vanderbilt, Nashville, Tennessee
  - MD Anderson, Houston, Texas
  - START, San Antonio, Texas
- Italy (2):
  - Ospedale San Raffaele, Milan
  - Oncologica Azienda Ospedaliera Universitaria Senese, Siena
- Netherlands (2):
  - NKI, Amsterdam
  - Radboudumc, Nijmegen
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Institut Catala d'Oncologia, Barcelona
  - START Madrid-HM CIOCC, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Naing A, Papadopoulos KP, Pishvaian MJ, Rahma O, Hanna GJ, Garralda E, Saavedra O, Gogov S, Kallender H, Cheng L, Smith M, Chen X, Kuriakose E, Bauer T. First-in-human phase 1 study of the arginase inhibitor INCB001158 alone or combined with pembrolizumab in patients with advanced or metastatic solid tumours. BMJ Oncol. 2024 May 9;3(1):e000249. doi: 10.1136/bmjonc-2023-000249. eCollection 2024. PMID 39886141
- [Derived] Aden D, Sureka N, Zaheer S, Chaurasia JK, Zaheer S. Metabolic Reprogramming in Cancer: Implications for Immunosuppressive Microenvironment. Immunology. 2025 Jan;174(1):30-72. doi: 10.1111/imm.13871. Epub 2024 Oct 27. PMID 39462179

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This global study (United States, Spain, and Italy) consisted of 3 parts: Part 1 was dose-escalation using a 3 + 3 design to determine the RP2D of INCB001158 as monotherapy (Part 1a) and in combination with pembrolizumab (Parts 1b and 1c); Part 2 and Part 3 consisted of tumor expansion cohorts to determine whether INCB001158 as monotherapy (Part 2) or in combination with pembrolizumab (Part 3) had sufficient antitumor activity and further evaluated the safety and tolerability of the RP2D.
Pre-assignment Details: 260 enrolled participants: 107 in the Part 1a and Part 2 monotherapy groups; 147 in the Part 1b and Part 3 combination therapy groups; and 6 in Part 1c. Disposition data have been reported by dose level; efficacy data have been reported by tumor type, regardless of dose received. One Part 3 participant scheduled to receive INCB001158 100 mg actually received 75 mg; they were included in the Part 1b 75 mg arm for disposition analysis and in the Part 1c and Part 3 100 mg arm for efficacy analysis.
Groups:
- Part 1A: INCB001158 50 mg: INCB001158 was administered orally at 50 milligrams (mg) twice daily (BID) in participants with advanced/metastatic solid tumors.
- Part 1A: INCB001158 75 mg: INCB001158 was administered orally at 75 mg BID in participants with advanced/metastatic solid tumors.
- Part 1A and Part 2: INCB001158 100 mg: INCB001158 was administered orally at 100 mg BID in participants with advanced/metastatic solid tumors.
- Part 1A: INCB001158 150 mg: INCB001158 was administered orally at 150 mg BID in participants with advanced/metastatic solid tumors.
- Part 1B: INCB001158 50 mg + Pembrolizumab: INCB001158 was administered orally at 50 mg BID in combination with pembrolizumab at 200 mg intravenously (IV) every 3 weeks (Q3W).
- Part 1B: INCB001158 75 mg + Pembrolizumab: INCB001158 was administered orally at 75 mg BID in combination with pembrolizumab at 200 mg IV Q3W.
- Part 1B and Part 3: INCB001158 100 mg + Pembrolizumab: INCB001158 was administered orally at 100 mg BID in combination with pembrolizumab at 200 mg IV Q3W.
- Part 1C: INCB001158 50 mg + Pembrolizumab: INCB001158 was administered orally at 50 mg BID in combination with pembrolizumab at 200 mg IV Q3W to participants with moderately impaired renal function.
Period: Overall Study
Arm/Group | Part 1A: INCB001158 50 mg | Part 1A: INCB001158 75 mg | Part 1A and Part 2: INCB001158 100 mg | Part 1A: INCB001158 150 mg | Part 1B: INCB001158 50 mg + Pembrolizumab | Part 1B: INCB001158 75 mg + Pembrolizumab | Part 1B and Part 3: INCB001158 100 mg + Pembrolizumab | Part 1C: INCB001158 50 mg + Pembrolizumab
Started | 8 | 7 | 85 | 7 | 10 | 14 | 123 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 8 | 7 | 85 | 7 | 10 | 14 | 123 | 6
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 28 | 0 | 1 | 2 | 12 | 0
Not completed — Progressive Disease | 1 | 0 | 4 | 0 | 0 | 0 | 2 | 0
Not completed — Death | 0 | 0 | 9 | 0 | 1 | 3 | 24 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Symptomatic Deterioration | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — New Cancer Therapy | 2 | 2 | 21 | 4 | 3 | 6 | 56 | 3
Not completed — Didn't Return to Site | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 0
Not completed — Entered/Referred to Hospice Care | 1 | 1 | 8 | 0 | 0 | 0 | 4 | 0
Not completed — Follow-up Did Not Occur | 0 | 1 | 1 | 0 | 2 | 0 | 8 | 0
Not completed — Systemic Treatment Options Necessary | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Consented to/Considered Other Clinical Study | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0
Not completed — Clinical Disease Progression | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Completed Follow-up Period | 0 | 0 | 6 | 2 | 1 | 0 | 9 | 1
Not completed — Taken off Treatment per Protocol | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Refused Further Treatment/Contact | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Discontinued per Sponsor/Participant Agreement | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1A: INCB001158 50 mg | Part 1A: INCB001158 75 mg | Part 1A and Part 2: INCB001158 100 mg | Part 1A: INCB001158 150 mg | Part 1B: INCB001158 50 mg + Pembrolizumab | Part 1B: INCB001158 75 mg + Pembrolizumab | Part 1B and Part 3: INCB001158 100 mg + Pembrolizumab | Part 1C: INCB001158 50 mg + Pembrolizumab | Total
Number analyzed (Participants) | 8 | 7 | 85 | 7 | 10 | 14 | 123 | 6 | 260
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (3.96) | 61.7 (6.10) | 61.4 (10.42) | 67.0 (8.12) | 58.7 (11.64) | 62.8 (10.81) | 59.7 (11.94) | 73.3 (7.69) | 60.9 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 39 | 4 | 6 | 3 | 43 | 3 | 109
  Male | 3 | 1 | 46 | 3 | 4 | 11 | 80 | 3 | 151
Race/Ethnicity, Customized [Number; unit: Participants]
  White or Causasian | 5 | 7 | 70 | 6 | 9 | 13 | 109 | 5 | 224
  Black or African American | 2 | 0 | 11 | 1 | 0 | 0 | 3 | 1 | 18
  Asian | 1 | 0 | 3 | 0 | 1 | 1 | 4 | 0 | 10
  American Indican/Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Captured as "Other" in Database | 0 | 0 | 1 | 0 | 0 | 0 | 6 | 0 | 7
  Missing | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 2 | 1 | 10 | 1 | 0 | 0 | 7 | 0 | 21
  Not Hispanic or Latino | 6 | 6 | 75 | 6 | 10 | 14 | 114 | 6 | 237
  Missing | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related, that occurred after a participant provided informed consent. Abnormal laboratory values or test results occurring after informed consent constituted AEs only if they induced clinical signs or symptoms, were considered clinically meaningful, required therapy (e.g., hematologic abnormality that required transfusion), or required changes in the study treatment(s). A TEAE was defined as any adverse event that started or worsened after the first dose of study drug.
Time Frame: up to study completion (up to approximately 3.5 years)
Population: Safety Population: all participants who received at least 1 dose of INCB001158 or pembrolizumab. Data collected through study completion have been reported.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1A: INCB001158 100 mg: INCB001158 administered orally at 100mg BID in participants with advanced/metastatic solid tumors.
Arm/Group | Part 1A: INCB001158 50 mg | Part 1A: INCB001158 75 mg | Part 1A: INCB001158 100 mg | Part 1A: INCB001158 150 mg | Part 1B: INCB001158 50 mg + Pembrolizumab | Part 1B: INCB001158 75 mg + Pembrolizumab | Part 1B and Part 3: INCB001158 100 mg + Pembrolizumab | Part 1C: INCB001158 50 mg + Pembrolizumab
Number analyzed (Participants) | 8 | 7 | 85 | 7 | 10 | 14 | 123 | 6
Participants | 7 | 7 | 81 | 7 | 10 | 13 | 123 | 6

2. Secondary Outcome: Recommended Phase 2 Dose (RP2D) of INCB001158
Description: The RP2D was determined by a traditional 3+3 dose-escalation design of single-agent INCB001158 in participants with advanced/metastatic solid tumors at doses of 50, 75, 100, or 150 mg.
Time Frame: 12 weeks
Population: Safety Population
Measure: Number; unit: milligrams
Groups:
- INCB001158 as Monotherapy at 50, 75, 100 and 150 mg BID: Monotherapy Part 1a: INCB001158 was administered orally in participants with advanced/metastatic solid tumors. Sequential dose escalation of single-agent INCB001158 took place in participants with advanced/metastatic solid tumors.
Arm/Group | INCB001158 as Monotherapy at 50, 75, 100 and 150 mg BID
Number analyzed (Participants) | 28
milligrams | 100

3. Secondary Outcome: RP2D of INCB001158 in Combination With Pembrolizumab
Description: INCB001158 was dosed orally BID.
Time Frame: 12 weeks
Population: Safety Population
Measure: Number; unit: milligrams
Groups:
- INCB001158 as Combination Therapy at 50, 75, and 100 mg BID: INCB001158 administered orally in patients at 50, 75, and 100 mg doses BID with advanced/metastatic solid tumors in combination with pembrolizumab (200 mg IV Q3W)
Arm/Group | INCB001158 as Combination Therapy at 50, 75, and 100 mg BID
Number analyzed (Participants) | 33
milligrams | 100

4. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (v1.1) as the percentage of participants with a confirmed best overall response of complete response (CR) or partial response (PR) at any post-Baseline visits prior to first disease progression and alternative cancer therapy use. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 millimeters (mm). PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions. Pleural mesothelioma was evaluated using modified RECIST criteria. Confidence intervals were calculated based on the exact method for binomial distributions (Clopper Pearson). Two participants evaluable for PFS were not evaluable for response.
Time Frame: Until disease progression/study discontinuation (up to approximately 5 years)
Population: Response Efficacy Evaluable Population (REEP): received ≥1 dose of INCB001158 or pembrolizumab, completed a Baseline scan, and met ≥1 protocol-defined criteria. Part 1c participants had renal impairment and received INCB001158 50 mg + pembrolizumab, which was half the recommended Phase 2 dose of INCB001158. It was pre-specified to combine Part 1c and Part 3 participants for efficacy analysis based on planned comparable dosing according to renal function.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part 1A: INCB001158 100 mg; Part 2: INCB001158 100 mg: INCB001158 was administered orally at 100 mg BID in participants with advanced/metastatic solid tumors.
- Part 1B: INCB001158 100 mg + Pembrolizumab: INCB001158 was administered orally at 100 mg BID in combination with pembrolizumab at 200 mg IV Q3W.
- Part 1c and Part 3: INCB001158 100 mg + Pembrolizumab: INCB001158 was administered orally at 100 mg BID (50 mg BID for Part 1c renally impaired participants) in combination with pembrolizumab at 200 mg IV Q3W.
Arm/Group | Part 1A: INCB001158 50 mg | Part 1A: INCB001158 75 mg | Part 1A: INCB001158 100 mg | Part 1A: INCB001158 150 mg | Part 1B: INCB001158 50 mg + Pembrolizumab | Part 1B: INCB001158 75 mg + Pembrolizumab | Part 1B: INCB001158 100 mg + Pembrolizumab | Part 2: INCB001158 100 mg | Part 1c and Part 3: INCB001158 100 mg + Pembrolizumab
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 10 | 13 | 10 | 73 | 118
percentage of participants | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 45.9] | 10.0 [0.3 to 44.5] | 7.7 [0.2 to 36.0] | 0.0 [0.0 to 30.8] | 1.4 [0.0 to 7.4] | 11.0 [6.0 to 18.1]

5. Secondary Outcome: Percentage of Participants With the Indicated Best Overall Response (BOR)
Description: BOR was evaluated per RECIST v1.1. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 mm. PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions. Stable disease (SD): no change in target lesions to qualify for CR, PR, or progressive disease (PD). PD: progression of a target or non-target lesion or presence of a new lesion. Missing: participant had a missing BOR because there were no post-Baseline tumor assessments. Pleural mesothelioma was evaluated using modified RECIST criteria.
Time Frame: Until disease progression/study discontinuation (up to approximately 5 years)
Population: REEP. Participants enrolled in Part 1c had renal impairment. These participants received INCB001158 50 mg + pembrolizumab, which was half the recommended Phase 2 dose of INCB001158. It was pre-specified to combine Part 1c and Part 3 participants for efficacy analysis based on planned comparable dosing according to renal function. Two participants evaluable for PFS were not evaluable for response.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1A: INCB001158 50 mg | Part 1A: INCB001158 75 mg | Part 1A: INCB001158 100 mg | Part 1A: INCB001158 150 mg | Part 1B: INCB001158 50 mg + Pembrolizumab | Part 1B: INCB001158 75 mg + Pembrolizumab | Part 1B: INCB001158 100 mg + Pembrolizumab | Part 2: INCB001158 100 mg | Part 1c and Part 3: INCB001158 100 mg + Pembrolizumab
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 10 | 13 | 10 | 73 | 118
percentage of participants
  Complete Response | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 1.7
  Partial Response | 0.0 | 0.0 | 0.0 | 0.0 | 10.0 | 7.7 | 0.0 | 1.4 | 9.3
  Stable Disease | 33.3 | 0.0 | 16.7 | 33.3 | 10.0 | 38.5 | 20.0 | 30.1 | 36.4
  Progressive Disease | 66.7 | 85.7 | 83.3 | 66.7 | 70.0 | 46.2 | 80.0 | 50.7 | 44.9
  Not Evaluable | 0.0 | 14.3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 4.1 | 4.2
  Not Assessed | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Missing | 0.0 | 0.0 | 0.0 | 0.0 | 10.0 | 7.7 | 0.0 | 13.7 | 3.4

6. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the number of months from the date of the first documentation of an objective response (CR or PR per RECIST v1.1) to the date of the first documentation of disease progression or death, whichever occurred first. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 millimeters (mm). PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions. Pleural mesothelioma will be evaluated using modified RECIST criteria. Kaplan-Meier (KM) product-limit estimates with a log-log transformation were used for 95% confidence interval calculation.
Time Frame: Until disease progression/study discontinuation (up to approximately 5 years)
Population: REEP. Only participants with CR or PR were analyzed, and only cohorts with ≥5 objective responders were analyzed. Part 1c participants had renal impairment and received INCB001158 50 mg + pembrolizumab (half the RP2D of INCB001158). It was pre-specified to combine Part 1c and Part 3 participants for efficacy analysis based on planned comparable dosing according to renal function. Two participants evaluable for PFS were not evaluable for response.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Part 1c and Part 3, SCCHN: INCB001158 100 mg + Pembrolizumab: INCB001158 was administered orally at 100 mg BID (50 mg BID for Part 1c renally impaired participants) in combination with pembrolizumab at 200 mg IV Q3W to participants with squamous cell carcinoma of the head and neck (SCCHN).
Arm/Group | Part 1A: INCB001158 50 mg | Part 1A: INCB001158 75 mg | Part 1A: INCB001158 100 mg | Part 1A: INCB001158 150 mg | Part 1B: INCB001158 50 mg + Pembrolizumab | Part 1B: INCB001158 75 mg + Pembrolizumab | Part 1B: INCB001158 100 mg + Pembrolizumab | Part 2: INCB001158 100 mg | Part 1c and Part 3, SCCHN: INCB001158 100 mg + Pembrolizumab
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 5
months |  |  |  |  | NA [NA to NA] — The KM estimation method on a sample of <5 responders is not valid because too few participants were responders. | NA [NA to NA] — The KM estimation method on a sample of <5 responders is not valid because too few participants were responders. |  | NA [NA to NA] — The KM estimation method on a sample of <5 responders is not valid because too few participants were responders. | 12.4 [4.2 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died.

7. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the length of time between the date of the first dose and the earlier of death or progressive disease as assessed by RECIST v1.1. Pleural mesothelioma was evaluated using modified RECIST criteria. Participants enrolled in Part 1c had renal impairment. These participants received INCB001158 50 mg + pembrolizumab, which was half the recommended Phase 2 dose of INCB001158. In renally impaired participants, the 50 mg dose has comparable exposure to 100 mg in participants with normal renal function. It was pre-specified to combine Part 1c and Part 3 participants for efficacy analysis based on planned comparable dosing according to renal function.
Time Frame: Until disease progression/study discontinuation (up to approximately 5 years)
Population: PFS Efficacy Evaluable Population (Full Analysis Set): all participants who received at least 1 dose of INCB001158 or pembrolizumab. One participant was to be treated with INCB001158 100 mg + pembrolizumab but actually received INCB001158 75 mg + pembrolizumab. For PFS analysis, this participant was analyzed in their planned treatment group (INCB001158 100 mg + pembrolizumab) rather than in the actual treatment group.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1A: INCB001158 50 mg | Part 1A: INCB001158 75 mg | Part 1A: INCB001158 100 mg | Part 1A: INCB001158 150 mg | Part 1B: INCB001158 50 mg + Pembrolizumab | Part 1B: INCB001158 75 mg + Pembrolizumab | Part 1B: INCB001158 100 mg + Pembrolizumab | Part 2: INCB001158 100 mg | Part 1c and Part 3: INCB001158 100 mg + Pembrolizumab
Number analyzed (Participants) | 8 | 7 | 8 | 7 | 10 | 13 | 11 | 77 | 119
months | 1.8 [1.2 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 1.8 [1.2 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 1.8 [1.4 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 2.1 [1.7 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 2.1 [0.7 to 6.2] | 2.6 [1.8 to 5.7] | 2.1 [0.6 to 2.3] | 1.9 [1.8 to 2.1] | 3.0 [2.1 to 4.1]

8. Secondary Outcome: Cmax of INCB001158 Following Single Escalating Doses for Part 1A
Description: Cmax was defined as the maximum observed concentration of INCB001158.
Time Frame: Cycle 1 Day 1: predose; 0.5, 1, 2, 4, 6, 8, 12, and 24 hours post-dose
Population: Pharmacokinetic (PK) Population: all participants who received at least 1 dose of INCB001158 or pembrolizumab and contributed at least 1 PK sample
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Part 1A: INCB001158 50 mg | Part 1A: INCB001158 75 mg | Part 1A: INCB001158 100 mg | Part 1A: INCB001158 150 mg
Number analyzed (Participants) | 8 | 7 | 8 | 7
nanograms per milliliter (ng/mL) | 763 (0.30) | 1310 (0.26) | 1420 (0.30) | 1990 (0.33)
Statistical Analysis 1: Comparison: Part 1A: INCB001158 50 mg vs Part 1A: INCB001158 75 mg vs Part 1A: INCB001158 100 mg vs Part 1A: INCB001158 150 mg; Test type: Other; p = 0.0731, ANOVA; 1-factor ANOVA of log-transformed, dose-normalized data (factor = dose)
Statistical Analysis 2: Comparison: Part 1A: INCB001158 100 mg vs Part 1A: INCB001158 150 mg; Test type: Other; pairwise geometric mean ratio (GMR) = 0.933, 90% CI 2-sided [0.784 to 1.110]
Statistical Analysis 3: Comparison: Part 1A: INCB001158 50 mg vs Part 1A: INCB001158 100 mg; Test type: Other; pairwise GMR = 1.074, 90% CI 2-sided [0.908 to 1.271]
Statistical Analysis 4: Comparison: Part 1A: INCB001158 75 mg vs Part 1A: INCB001158 100 mg; Test type: Other; pairwise GMR = 1.230, 90% CI 2-sided [1.034 to 1.463]

9. Secondary Outcome: Tmax of INCB001158 Following Single Escalating Doses for Part 1A
Description: tmax was defined as the time of the maximum observed concentration of INCB001158.
Time Frame: Cycle 1 Day 1: predose; 0.5, 1, 2, 4, 6, 8, 12, and 24 hours post-dose
Population: PK Population
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1A: INCB001158 50 mg | Part 1A: INCB001158 75 mg | Part 1A: INCB001158 100 mg | Part 1A: INCB001158 150 mg
Number analyzed (Participants) | 8 | 7 | 8 | 7
hours | 3.9 [2.0 to 4.1] | 2.0 [2.0 to 6.2] | 4.0 [2.1 to 6.1] | 6.0 [3.8 to 6.0]
Statistical Analysis 1: Comparison: Part 1A: INCB001158 50 mg vs Part 1A: INCB001158 75 mg vs Part 1A: INCB001158 100 mg vs Part 1A: INCB001158 150 mg; Test type: Other; p = 0.1496, Kruskal-Wallis; 1-factor ANOVA of log-transformed, dose-normalized data (factor = dose)

10. Secondary Outcome: AUC0-t of INCB001158 Following Single Escalating Doses for Part 1A
Description: AUC0-t was defined as the area under the concentration-time curve from dosing (time 0) of INCB001158 to time t.
Time Frame: Cycle 1 Day 1: predose; 0.5, 1, 2, 4, 6, 8, 12, and 24 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours x ng/mL
Arm/Group | Part 1A: INCB001158 50 mg | Part 1A: INCB001158 75 mg | Part 1A: INCB001158 100 mg | Part 1A: INCB001158 150 mg
Number analyzed (Participants) | 8 | 7 | 8 | 7
hours x ng/mL | 7700 (0.32) | 13200 (0.34) | 14200 (0.37) | 21500 (0.35)
Statistical Analysis 1: Comparison: Part 1A: INCB001158 50 mg vs Part 1A: INCB001158 75 mg vs Part 1A: INCB001158 100 mg vs Part 1A: INCB001158 150 mg; Test type: Other; p = 0.2867, ANOVA; 1-factor ANOVA of log-transformed, dose-normalized data (factor = dose)
Statistical Analysis 2: Comparison: Part 1A: INCB001158 100 mg vs Part 1A: INCB001158 150 mg; Test type: Other; pairwise GMR = 1.007, 90% CI 2-sided [0.825 to 1.230]
Statistical Analysis 3: Comparison: Part 1A: INCB001158 50 mg vs Part 1A: INCB001158 100 mg; Test type: Other; pairwise GMR = 1.081, 90% CI 2-sided [0.892 to 1.311]
Statistical Analysis 4: Comparison: Part 1A: INCB001158 75 mg vs Part 1A: INCB001158 100 mg; Test type: Other; pairwise GMR = 1.234, 90% CI 2-sided [1.011 to 1.507]

11. Secondary Outcome: AUC0-inf of INCB001158 Following Single Escalating Doses for Part 1A
Description: AUC0-inf was defined as the area under the concentration-time curve from dosing (time 0) of INCB001158 extrapolated to infinity.
Time Frame: Cycle 1 Day 1: predose; 0.5, 1, 2, 4, 6, 8, 12, and 24 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours x ng/mL
Arm/Group | Part 1A: INCB001158 50 mg | Part 1A: INCB001158 75 mg | Part 1A: INCB001158 100 mg | Part 1A: INCB001158 150 mg
Number analyzed (Participants) | 8 | 7 | 8 | 7
hours x ng/mL | 8360 (0.35) | 14100 (0.38) | 16000 (0.42) | 24400 (0.34)
Statistical Analysis 1: Comparison: Part 1A: INCB001158 50 mg vs Part 1A: INCB001158 75 mg vs Part 1A: INCB001158 100 mg vs Part 1A: INCB001158 150 mg; Test type: Other; p = 0.6167, ANOVA; 1-factor ANOVA of log-transformed, dose-normalized data (factor = dose)
Statistical Analysis 2: Comparison: Part 1A: INCB001158 100 mg vs Part 1A: INCB001158 150 mg; Test type: Other; pairwise GMR = 1.014, 90% CI 2-sided [0.820 to 1.255]
Statistical Analysis 3: Comparison: Part 1A: INCB001158 50 mg vs Part 1A: INCB001158 100 mg; Test type: Other; pairwise GMR = 1.043, 90% CI 2-sided [0.849 to 1.281]
Statistical Analysis 4: Comparison: Part 1A: INCB001158 75 mg vs Part 1A: INCB001158 100 mg; Test type: Other; pairwise GMR = 1.170, 90% CI 2-sided [0.945 to 1.447]

12. Secondary Outcome: t1/2 of INCB001158 Following Single Escalating Doses for Part 1A
Description: t1/2 was defined as the half-life of INCB001158.
Time Frame: Cycle 1 Day 1: predose; 0.5, 1, 2, 4, 6, 8, 12, and 24 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 1A: INCB001158 50 mg | Part 1A: INCB001158 75 mg | Part 1A: INCB001158 100 mg | Part 1A: INCB001158 150 mg
Number analyzed (Participants) | 8 | 7 | 8 | 7
hours | 5.33 (0.25) | 5.21 (0.17) | 5.70 (0.13) | 5.65 (0.15)

13. Secondary Outcome: CL/F of INCB001158 Following Single Escalating Doses for Part 1A
Description: CL/F was defined as the apparent oral dose clearance of INCB001158.
Time Frame: Cycle 1 Day 1: predose; 0.5, 1, 2, 4, 6, 8, 12, and 24 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Part 1A: INCB001158 50 mg | Part 1A: INCB001158 75 mg | Part 1A: INCB001158 100 mg | Part 1A: INCB001158 150 mg
Number analyzed (Participants) | 8 | 7 | 8 | 7
Liters per hour | 5980 (0.35) | 5330 (0.38) | 6240 (0.42) | 6150 (0.34)

14. Secondary Outcome: Vz/F of INCB001158 Following Single Escalating Doses for Part 1A
Description: Vz/F was defined as the apparent volume of distribution of INCB001158.
Time Frame: Cycle 1 Day 1: predose; 0.5, 1, 2, 4, 6, 8, 12, and 24 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Part 1A: INCB001158 50 mg | Part 1A: INCB001158 75 mg | Part 1A: INCB001158 100 mg | Part 1A: INCB001158 150 mg
Number analyzed (Participants) | 8 | 7 | 8 | 7
Liters | 46000 (0.29) | 40100 (0.22) | 51300 (0.32) | 50100 (0.30)

15. Secondary Outcome: Cmax of INCB001158 Following Multiple Escalating Doses for Part 1A
Description: Cmax was defined as the maximum observed concentration of INCB001158.
Time Frame: Cycle 1 Day 15: predose; 0.5, 1, 2, 4, 6, 8, and 12 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1A: INCB001158 50 mg | Part 1A: INCB001158 75 mg | Part 1A: INCB001158 100 mg | Part 1A: INCB001158 150 mg
Number analyzed (Participants) | 6 | 7 | 7 | 6
ng/mL | 987 (0.28) | 1880 (0.28) | 1990 (0.26) | 3370 (0.30)
Statistical Analysis 1: Comparison: Part 1A: INCB001158 50 mg vs Part 1A: INCB001158 75 mg vs Part 1A: INCB001158 100 mg vs Part 1A: INCB001158 150 mg; Test type: Other; p = 0.0745, ANOVA; 1-factor ANOVA of log-transformed, dose-normalized data (factor = dose)
Statistical Analysis 2: Comparison: Part 1A: INCB001158 100 mg vs Part 1A: INCB001158 150 mg; Test type: Other; pairwise GMR = 1.127, 90% CI 2-sided [0.947 to 1.341]
Statistical Analysis 3: Comparison: Part 1A: INCB001158 50 mg vs Part 1A: INCB001158 100 mg; Test type: Other; pairwise GMR = 0.991, 90% CI 2-sided [0.833 to 1.180]
Statistical Analysis 4: Comparison: Part 1A: INCB001158 75 mg vs Part 1A: INCB001158 100 mg; Test type: Other; pairwise GMR = 1.258, 90% CI 2-sided [1.064 to 1.486]

16. Secondary Outcome: Tmax of INCB001158 Following Multiple Escalating Doses for Part 1A
Description: tmax was defined as the time of the maximum observed concentration of INCB001158.
Time Frame: Cycle 1 Day 15: predose; 0.5, 1, 2, 4, 6, 8, and 12 hours post-dose
Population: PK Population
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1A: INCB001158 50 mg | Part 1A: INCB001158 75 mg | Part 1A: INCB001158 100 mg | Part 1A: INCB001158 150 mg
Number analyzed (Participants) | 6 | 7 | 7 | 6
hours | 2.0 [1.9 to 4.0] | 4.1 [2.0 to 6.1] | 4.0 [2.1 to 5.9] | 2.0 [1.9 to 4.2]
Statistical Analysis 1: Comparison: Part 1A: INCB001158 50 mg vs Part 1A: INCB001158 75 mg vs Part 1A: INCB001158 100 mg vs Part 1A: INCB001158 150 mg; Test type: Other; p = 0.0518, Kruskal-Wallis

17. Secondary Outcome: AUC0-t of INCB001158 Following Multiple Escalating Doses for Part 1A
Description: AUC0-t was defined as the area under the concentration-time curve from dosing (time 0) of INCB001158 to time t.
Time Frame: Cycle 1 Day 15: predose; 0.5, 1, 2, 4, 6, 8, and 12 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours x ng/mL
Arm/Group | Part 1A: INCB001158 50 mg | Part 1A: INCB001158 75 mg | Part 1A: INCB001158 100 mg | Part 1A: INCB001158 150 mg
Number analyzed (Participants) | 6 | 7 | 7 | 6
hours x ng/mL | 7910 (0.26) | 15000 (0.35) | 16200 (0.38) | 28100 (0.32)
Statistical Analysis 1: Comparison: Part 1A: INCB001158 50 mg vs Part 1A: INCB001158 75 mg vs Part 1A: INCB001158 100 mg vs Part 1A: INCB001158 150 mg; Test type: Other; p = 0.1723, ANOVA; 1-factor ANOVA of log-transformed, dose-normalized data (factor = dose)
Statistical Analysis 2: Comparison: Part 1A: INCB001158 100 mg vs Part 1A: INCB001158 150 mg; Test type: Other; pairwise GMR = 1.156, 90% CI 2-sided [0.941 to 1.420]
Statistical Analysis 3: Comparison: Part 1A: INCB001158 50 mg vs Part 1A: INCB001158 100 mg; Test type: Other; pairwise GMR = 0.976, 90% CI 2-sided [0.794 to 1.198]
Statistical Analysis 4: Comparison: Part 1A: INCB001158 75 mg vs Part 1A: INCB001158 100 mg; Test type: Other; pairwise GMR = 1.233, 90% CI 2-sided [1.012 to 1.503]

18. Secondary Outcome: AUC0-tau of INCB001158 Following Multiple Escalating Doses for Part 1A
Description: AUC0-tau was defined as the area under the concentration-time curve from dosing (time 0) of INCB001158 to the end of the dosing period.
Time Frame: Cycle 1 Day 15: predose; 0.5, 1, 2, 4, 6, 8, and 12 hours post-dose
Population: PK Population. Only participants with available data were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours x ng/mL
Arm/Group | Part 1A: INCB001158 50 mg | Part 1A: INCB001158 75 mg | Part 1A: INCB001158 100 mg | Part 1A: INCB001158 150 mg
Number analyzed (Participants) | 6 | 4 | 4 | 6
hours x ng/mL | 8250 (0.27) | 16600 (0.39) | 18300 (0.34) | 29700 (0.31)
Statistical Analysis 1: Comparison: Part 1A: INCB001158 50 mg vs Part 1A: INCB001158 75 mg vs Part 1A: INCB001158 100 mg vs Part 1A: INCB001158 150 mg; Test type: Other; p = 0.1705, ANOVA; 1-factor ANOVA of log-transformed, dose-normalized data (factor = dose)
Statistical Analysis 2: Comparison: Part 1A: INCB001158 100 mg vs Part 1A: INCB001158 150 mg; Test type: Other; pairwise GMR = 1.083, 90% CI 2-sided [0.863 to 1.359]
Statistical Analysis 3: Comparison: Part 1A: INCB001158 50 mg vs Part 1A: INCB001158 100 mg; Test type: Other; pairwise GMR = 0.902, 90% CI 2-sided [0.719 to 1.132]
Statistical Analysis 4: Comparison: Part 1A: INCB001158 75 mg vs Part 1A: INCB001158 100 mg; Test type: Other; pairwise GMR = 1.212, 90% CI 2-sided [0.945 to 1.554]

19. Secondary Outcome: t1/2 of INCB001158 Following Multiple Escalating Doses for Part 1A
Description: t1/2 was defined as the half-life of INCB001158.
Time Frame: Cycle 1 Day 15: predose; 0.5, 1, 2, 4, 6, 8, and 12 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 1A: INCB001158 50 mg | Part 1A: INCB001158 75 mg | Part 1A: INCB001158 100 mg | Part 1A: INCB001158 150 mg
Number analyzed (Participants) | 6 | 4 | 4 | 6
hours | 5.54 (0.22) | 5.22 (0.22) | 5.70 (0.40) | 6.83 (0.28)

20. Secondary Outcome: CL/F of INCB001158 Following Multiple Escalating Doses for Part 1A
Description: CL/F was defined as the apparent oral dose clearance of INCB001158.
Time Frame: Cycle 1 Day 15: predose; 0.5, 1, 2, 4, 6, 8, and 12 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Part 1A: INCB001158 50 mg | Part 1A: INCB001158 75 mg | Part 1A: INCB001158 100 mg | Part 1A: INCB001158 150 mg
Number analyzed (Participants) | 6 | 4 | 4 | 6
Liters per hour | 6060 (0.27) | 4510 (0.39) | 5470 (0.34) | 5050 (0.31)

21. Secondary Outcome: Vz/F of INCB001158 Following Multiple Escalating Doses for Part 1A
Description: Vz/F was defined as the apparent volume of distribution of INCB001158.
Time Frame: Cycle 1 Day 15: predose; 0.5, 1, 2, 4, 6, 8, and 12 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Part 1A: INCB001158 50 mg | Part 1A: INCB001158 75 mg | Part 1A: INCB001158 100 mg | Part 1A: INCB001158 150 mg
Number analyzed (Participants) | 6 | 4 | 4 | 6
Liters | 48400 (0.34) | 34000 (0.48) | 45000 (0.09) | 49700 (0.30)

22. Secondary Outcome: Cmax of INCB001158 in the Fed and Fasted States Following Multiple Doses for Part 1A to Assess the Effect of Food
Description: Cmax was defined as the maximum observed concentration of INCB001158.
Time Frame: Fasted: Cycle 1 Day 15: predose; 0.5, 1, 2, 4, 6, 8, and 12 hours post-dose. Fed: Cycle 2 Day 8: predose; 0.5, 1, 2, 4, 6, and 8 hours post-dose
Population: PK Population. Only participants with available date were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1A: INCB001158 50 mg | Part 1A: INCB001158 75 mg | Part 1A: INCB001158 100 mg | Part 1A: INCB001158 150 mg
Number analyzed (Participants) | 6 | 7 | 7 | 6
ng/mL
  Fasted: number analyzed (Participants) | 5 | 5 | 7 | 6
  Fasted | 904 (0.19) | 1840 (0.31) | 1990 (0.26) | 3370 (0.30)
  Fed: number analyzed (Participants) | 6 | 6 | 6 | 3
  Fed | 955 (0.38) | 1860 (0.22) | 2130 (0.31) | 4170 (0.32)
Statistical Analysis 1: Comparison: Part 1A: INCB001158 50 mg; Fed versus Fasted; Test type: Other; p = 0.7702, ANOVA; 1-factor ANOVA of log-transformed, dose-normalized data (factor = food effect); pairwise GMR = 1.057, 90% CI 2-sided [0.753 to 1.483]
Statistical Analysis 2: Comparison: Part 1A: INCB001158 75 mg; Fed versus Fasted; Test type: Other; p = 0.9384, ANOVA; 1-factor ANOVA of log-transformed, dose-normalized data (factor = food effect); pairwise GMR = 1.012, 90% CI 2-sided [0.762 to 1.346]
Statistical Analysis 3: Comparison: Part 1A: INCB001158 100 mg; Fed versus Fasted; Test type: Other; p = 0.6733, ANOVA; 1-factor ANOVA of log-transformed, dose-normalized data (factor = food effect); pairwise GMR = 1.070, 90% CI 2-sided [0.809 to 1.415]
Statistical Analysis 4: Comparison: Part 1A: INCB001158 150 mg; Fed versus Fasted; Test type: Other; p = 0.3456, ANOVA; 1-factor ANOVA of log-transformed, dose-normalized data (factor = food effect); pairwise GMR = 1.238, 90% CI 2-sided [0.830 to 1.847]

23. Secondary Outcome: Tmax of INCB001158 in the Fed and Fasted States Following Multiple Doses for Part 1A to Assess the Effect of Food
Description: tmax was defined as the time of the maximum observed concentration of INCB001158.
Time Frame: as for outcome 22
Population: PK Population. Only participants with available data were analyzed.
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1A: INCB001158 50 mg | Part 1A: INCB001158 75 mg | Part 1A: INCB001158 100 mg | Part 1A: INCB001158 150 mg
Number analyzed (Participants) | 6 | 7 | 7 | 6
hours
  Fasted | 2.0 [2.0 to 4.0] | 4.0 [2.0 to 4.3] | 4.0 [2.1 to 5.9] | 2.0 [1.9 to 4.2]
  Fed: number analyzed (Participants) | 6 | 6 | 6 | 3
  Fed | 4.0 [3.9 to 7.2] | 4.0 [4.0 to 6.1] | 4.0 [3.8 to 6.0] | 4.0 [4.0 to 6.2]
Statistical Analysis 1: Comparison: Part 1A: INCB001158 50 mg; Fed versus Fasted; Test type: Other; p = 0.0441, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Part 1A: INCB001158 75 mg; Fed versus Fasted; Test type: Other; p = 0.4092, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Part 1A: INCB001158 100 mg; Fed versus Fasted; Test type: Other; p = 0.7748, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Part 1A: INCB001158 150 mg; Fed versus Fasted; Test type: Other; p = 0.1948, Wilcoxon (Mann-Whitney)

24. Secondary Outcome: AUC of INCB001158 in the Fed and Fasted States Following Multiple Doses for Part 1A to Assess the Effect of Food
Description: AUC was defined as the area under the concentration-time curve of INCB001158.
Time Frame: as for outcome 22
Population: PK Population. Only participants with available date were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours x ng/mL
Arm/Group | Part 1A: INCB001158 50 mg | Part 1A: INCB001158 75 mg | Part 1A: INCB001158 100 mg | Part 1A: INCB001158 150 mg
Number analyzed (Participants) | 6 | 7 | 7 | 6
hours x ng/mL
  Fasted: number analyzed (Participants) | 5 | 5 | 7 | 6
  Fasted | 6030 (0.26) | 11900 (0.37) | 13100 (0.31) | 22100 (0.29)
  Fed: number analyzed (Participants) | 6 | 6 | 6 | 3
  Fed | 55550 (0.44) | 11000 (0.27) | 13100 (0.35) | 16400 (0.89)
Statistical Analysis 1: Comparison: Part 1A: INCB001158 50 mg; Fed versus Fasted; Test type: Other; p = 0.7050, ANOVA; 1-factor ANOVA of log-transformed, dose-normalized data (factor = food effect); pairwise GMR = 0.920, 90% CI 2-sided [0.620 to 1.363]
Statistical Analysis 2: Comparison: Part 1A: INCB001158 75 mg; Fed versus Fasted; Test type: Other; p = 0.7030, ANOVA; 1-factor ANOVA of log-transformed, dose-normalized data (factor = food effect); pairwise GMR = 0.929, 90% CI 2-sided [0.658 to 1.310]
Statistical Analysis 3: Comparison: Part 1A: INCB001158 100 mg; Fed versus Fasted; Test type: Other; p = 0.9952, ANOVA; 1-factor ANOVA of log-transformed, dose-normalized data (factor = food effect); pairwise GMR = 0.999, 90% CI 2-sided [0.725 to 1.377]
Statistical Analysis 4: Comparison: Part 1A: INCB001158 150 mg; Fed versus Fasted; Test type: Other; p = 0.4012, ANOVA; 1-factor ANOVA of log-transformed, dose-normalized data (factor = food effect); pairwise GMR = 0.742, 90% CI 2-sided [0.394 to 1.397]

25. Secondary Outcome: Cmax of INCB001158 for Capsules Versus Tablets for Part 2D to Assess the Effect of Formulation
Description: Cmax was defined as the maximum observed concentration of INCB001158.
Time Frame: Tablet: Cycle 1 Day 15 (Tablet) and Cycle 2 Day 1 (Capsule): predose; 0.5, 1, 2, 4, 6, 8, and 10 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part 2D: INCB001158 100 mg: INCB001158 was administered orally at 100 mg BID in participants with advanced/metastatic solid tumors. Participants enrolled in Part 2D received INCB001158 tablets from C1D1 to C1D15, and then switched to INCB001158 capsules starting on C1D16 onwards.
Arm/Group | Part 2D: INCB001158 100 mg
Number analyzed (Participants) | 5
ng/mL
  Capsule | 2170 (0.23)
  Tablet | 2150 (0.29)
Statistical Analysis 1: Comparison: Part 2D: INCB001158 100 mg; Tablet (test) versus Capsule (reference); Test type: Other; p = 0.9623, ANOVA; 1-factor ANOVA of log-transformed, dose-normalized data (factor = formulation); pairwise GMR = 0.992, 90% CI 2-sided [0.729 to 1.349]

26. Secondary Outcome: Tmax of INCB001158 for Capsules Versus Tablets for Part 2D to Assess the Effect of Formulation
Description: tmax was defined as the time of the maximum observed concentration of INCB001158.
Time Frame: Tablet: Cycle 1 Day 15 (Tablet) and Cycle 2 Day 1 (Capsule): predose; 0.5, 1, 2, 4, 6, 8, and 10 hours post-dose
Population: PK Population
Measure: Median (Full Range); unit: hours
Arm/Group | Part 2D: INCB001158 100 mg
Number analyzed (Participants) | 5
hours
  Capsule | 3.8 [1.8 to 6.0]
  Tablet | 3.8 [1.9 to 4.0]
Statistical Analysis 1: Comparison: Part 2D: INCB001158 100 mg; Tablet (test) versus Capsule (reference); Test type: Other; p = 0.7540, Wilcoxon (Mann-Whitney)

27. Secondary Outcome: AUC0-t of INCB001158 for Capsules Versus Tablets for Part 2D to Assess the Effect of Formulation
Description: AUC0-t was defined as the area under the concentration-time curve from dosing (time 0) of INCB001158 to time t.
Time Frame: Tablet: Cycle 1 Day 15 (Tablet) and Cycle 2 Day 1 (Capsule): predose; 0.5, 1, 2, 4, 6, 8, and 10 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours x ng/mL
Arm/Group | Part 2D: INCB001158 100 mg
Number analyzed (Participants) | 5
hours x ng/mL
  Capsule | 20800 (0.22)
  Tablet | 19700 (0.27)
Statistical Analysis 1: Comparison: Part 2D: INCB001158 100 mg; Tablet (test) versus Capsule (reference); Test type: Other; p = 0.7514, ANOVA; 1-factor ANOVA of log-transformed, dose-normalized data (factor = dose); pairwise GMR = 0.951, 90% CI 2-sided [0.718 to 1.261]

28. Secondary Outcome: AUC0-tau of INCB001158 for Capsules Versus Tablets for Part 2D to Assess the Effect of Formulation
Description: as for outcome 18
Time Frame: Tablet: Cycle 1 Day 15 (Tablet) and Cycle 2 Day 1 (Capsule): predose; 0.5, 1, 2, 4, 6, 8, and 10 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours x ng/mL
Arm/Group | Part 2D: INCB001158 100 mg
Number analyzed (Participants) | 5
hours x ng/mL
  Capsule | 18000 (0.22)
  Tablet | 17200 (0.28)
Statistical Analysis 1: Comparison: Part 2D: INCB001158 100 mg; Tablet (test) versus Capsule (reference); Test type: Other; p = 0.7707, ANOVA; 1-factor ANOVA of log-transformed, dose-normalized data (factor = formulation); pairwise GMR = 0.954, 90% CI 2-sided [0.712 to 1.277]

29. Secondary Outcome: Cmax of INCB001158 in Participants With Renal Impairment (Part 1C) and Normal Renal Function (Part 1A)
Description: Cmax was defined as the Maximum observed concentration of INCB001158.
Time Frame: Cycle 1 Day 1: predose; 0.5, 1, 2, 4, 6, 8, 12, and 24 (Part 1A only) hours post-dose.
Population: PK Population. Analysis was conducted to compare INCB001158 50 mg + pembrolizumab in participants with renal impairment with INCB001158 50 mg or 75 mg in participants with normal renal function. It was pre-specified to collect data for only the Part 1A INCB001158 50 mg, Part 1A: INCB001158 75 mg, and Part 1C: INCB001158 50 mg + Pembrolizumab arms. Participants in the INCB001158 100 mg and 150 mg arms did not contribute to the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1A: INCB001158 50 mg | Part 1A: INCB001158 75 mg | Part 1A: INCB001158 100 mg | Part 1A: INCB001158 150 mg | Part 1C: INCB001158 50 mg + Pembrolizumab
Number analyzed (Participants) | 8 | 7 | 0 | 0 | 6
ng/mL | 763 (0.30) | 1310 (0.26) |  |  | 1030 (0.21)

30. Secondary Outcome: Tmax of INCB001158 in Participants With Renal Impairment (Part 1C) and Normal Renal Function (Part 1A)
Description: tmax was defined as the time of the maximum observed concentration of INCB001158.
Time Frame: Cycle 1 Day 1: predose; 0.5, 1, 2, 4, 6, 8, 12, and 24 (Part 1A only) hours post-dose.
Population: as for outcome 29
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1A: INCB001158 50 mg | Part 1A: INCB001158 75 mg | Part 1A: INCB001158 100 mg | Part 1A: INCB001158 150 mg | Part 1C: INCB001158 50 mg + Pembrolizumab
Number analyzed (Participants) | 8 | 7 | 0 | 0 | 6
hours | 3.9 [2.0 to 4.1] | 2.0 [2.0 to 6.2] |  |  | 5.9 [3.9 to 7.9]

31. Secondary Outcome: AUC0-8h of INCB001158 in Participants With Renal Impairment (Part 1C) and Normal Renal Function (Part 1A)
Description: AUC0-8h was defined as the area under the concentration-time curve from dosing (time 0) of INCB001158 to 8 hours post-dose.
Time Frame: Cycle 1 Day 1: predose; 0.5, 1, 2, 4, 6, and 8 hours post-dose
Population: PK Population. Only participants with available data were analyzed. Analysis was conducted to compare INCB001158 50 mg + pembrolizumab in participants with renal impairment with INCB001158 50 mg or 75 mg in participants with normal renal function. It was pre-specified to collect data for only the Part 1A INCB001158 50 mg, Part 1A: INCB001158 75 mg, and Part 1C: INCB001158 50 mg + Pembrolizumab arms. Participants in the INCB001158 100 mg and 150 mg arms did not contribute to the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours x ng/mL
Arm/Group | Part 1A: INCB001158 50 mg | Part 1A: INCB001158 75 mg | Part 1A: INCB001158 100 mg | Part 1A: INCB001158 150 mg | Part 1C: INCB001158 50 mg + Pembrolizumab
Number analyzed (Participants) | 8 | 7 | 0 | 0 | 5
hours x ng/mL | 4480 (0.29) | 7890 (0.26) |  |  | 5210 (0.29)

ADVERSE EVENTS:
Time Frame: up to approximately 3.5 years
Description: For Adverse Event reporting, the data from Part 1C has been combined with that of Part 1B participants who received 50 mg INCB001158 + pembrolizumab.
Groups:
- Part 1B and Part 1C: INCB001158 50 mg + Pembrolizumab: INCB001158 was administered orally at 50 mg BID in combination with pembrolizumab at 200 mg intravenously (IV) every 3 weeks (Q3W). Participants in Part 1C had moderately impaired renal function.
- Total: Total
Arm/Group | Part 1A: INCB001158 50 mg | Part 1A: INCB001158 75 mg | Part 1A and Part 2: INCB001158 100 mg | Part 1A: INCB001158 150 mg | Part 1B and Part 1C: INCB001158 50 mg + Pembrolizumab | Part 1B: INCB001158 75 mg + Pembrolizumab | Part 1B and Part 3: INCB001158 100 mg + Pembrolizumab | Total
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7 | 12/85 | 0/7 | 3/16 | 3/14 | 24/123 | 42/260
Serious Adverse Events (participants affected / at risk) | 3/8 | 2/7 | 31/85 | 0/7 | 6/16 | 5/14 | 47/123 | 94/260
Other Adverse Events (participants affected / at risk) | 7/8 | 7/7 | 77/85 | 7/7 | 16/16 | 13/14 | 116/123 | 243/260
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1A: INCB001158 50 mg (N=8) | Part 1A: INCB001158 75 mg (N=7) | Part 1A and Part 2: INCB001158 100 mg (N=85) | Part 1A: INCB001158 150 mg (N=7) | Part 1B and Part 1C: INCB001158 50 mg + Pembrolizumab (N=16) | Part 1B: INCB001158 75 mg + Pembrolizumab (N=14) | Part 1B and Part 3: INCB001158 100 mg + Pembrolizumab (N=123) | Total (N=260)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 10 (13)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Adrenal haemorrhage (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Asymptomatic bacteriuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 6 (6)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 4 (4)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 4 (5)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 4 (5)
Empyema (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 6 (7)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (3)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 2 (2) | 3 (3) | 16 (16) | 26 (26)
Medical device site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 5 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (9) | 6 (10)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 5 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (3)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 4 (5)
Respirovirus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (5)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 6 (8)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1A: INCB001158 50 mg (N=8) | Part 1A: INCB001158 75 mg (N=7) | Part 1A and Part 2: INCB001158 100 mg (N=85) | Part 1A: INCB001158 150 mg (N=7) | Part 1B and Part 1C: INCB001158 50 mg + Pembrolizumab (N=16) | Part 1B: INCB001158 75 mg + Pembrolizumab (N=14) | Part 1B and Part 3: INCB001158 100 mg + Pembrolizumab (N=123) | Total (N=260)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 10 (10)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 11 (11) | 1 (1) | 2 (3) | 0 (0) | 3 (3) | 18 (19)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 6 (6)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 7 (8) | 9 (10)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 2 (2) | 21 (25) | 29 (33)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 3 (4) | 10 (11) | 0 (0) | 2 (2) | 1 (1) | 22 (23) | 41 (45)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 6 (6)
Appetite disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 11 (12) | 2 (3) | 0 (0) | 2 (2) | 14 (21) | 30 (39)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 7 (9) | 1 (1) | 1 (1) | 3 (3) | 23 (26) | 36 (41)
Asthenia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 11 (12) | 15 (16)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 8 (8) | 3 (4) | 0 (0) | 3 (3) | 15 (16) | 29 (31)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 12 (12) | 21 (21)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 9 (10) | 12 (13)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 8 (9) | 2 (2) | 0 (0) | 1 (1) | 17 (21) | 28 (33)
Blood iron decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (14) | 7 (14)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Breast tenderness (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (6)
Chills (General disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 8 (8) | 12 (12)
Cognitive disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 5 (6)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 18 (22) | 2 (2) | 0 (0) | 1 (1) | 29 (32) | 53 (60)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 7 (7) | 1 (1) | 1 (1) | 1 (1) | 16 (19) | 27 (30)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 17 (17) | 2 (2) | 3 (3) | 2 (2) | 22 (27) | 48 (53)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 6 (6) | 11 (12)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 4 (4) | 2 (2) | 31 (44) | 43 (56)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 13 (13) | 20 (21)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 1 (1) | 6 (6) | 13 (13)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 9 (9)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 8 (8) | 10 (10)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 12 (12) | 0 (0) | 1 (1) | 2 (2) | 16 (16) | 33 (33)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 7 (7)
Fatigue (General disorders) | 1 (1) | 3 (3) | 22 (23) | 3 (3) | 6 (6) | 3 (3) | 29 (31) | 67 (70)
Feeling abnormal (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 5 (5)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 5 (5)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 6 (7)
Haematochezia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 10 (14) | 17 (21)
Haemorrhoids (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 6 (6) | 0 (0) | 0 (0) | 1 (1) | 7 (10) | 15 (18)
Hepatobiliary disease (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 8 (8)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 3 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 7 (12) | 1 (1) | 1 (1) | 1 (2) | 7 (9) | 18 (26)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 6 (7)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 7 (7)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 6 (8) | 1 (1) | 0 (0) | 2 (2) | 22 (33) | 31 (44)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 5 (6)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 12 (15) | 12 (15)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 12 (15) | 15 (18)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 3 (3) | 28 (35) | 36 (43)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 11 (17) | 15 (21)
Hypotension (Vascular disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 8 (9)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 3 (4) | 13 (16) | 20 (24)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 4 (4)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 9 (10) | 19 (20)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 5 (5)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Local swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Metamorphopsia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (3) | 1 (2) | 0 (0) | 1 (1) | 2 (3) | 7 (10)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 8 (8)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 11 (11)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 6 (7) | 2 (2) | 1 (1) | 1 (1) | 6 (6) | 16 (17)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 10 (10) | 14 (14)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (3) | 3 (4) | 18 (21) | 1 (2) | 3 (3) | 0 (0) | 22 (25) | 49 (58)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 4 (7) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 11 (14)
Nodule (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Oedema peripheral (General disorders) | 2 (3) | 0 (0) | 12 (12) | 1 (1) | 1 (1) | 3 (4) | 8 (9) | 27 (30)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 6 (6)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 7 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 6 (6) | 1 (1) | 0 (0) | 3 (5) | 4 (4) | 15 (17)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Paraesthesia oral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 6 (6)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 4 (4)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 2 (2) | 1 (1) | 6 (7)
Procedural pain (General disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (12) | 7 (13)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 9 (9) | 12 (12)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 4 (5) | 2 (2) | 0 (0) | 0 (0) | 14 (18) | 22 (27)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 11 (11) | 16 (17)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (6) | 7 (7)
Renal vein thrombosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 5 (5)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stoma site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 2 (3)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 5 (6)
Temperature intolerance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 7 (7) | 9 (9)
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 8 (10) | 12 (14)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (4) | 2 (2) | 2 (3) | 0 (0) | 9 (13) | 16 (22)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Visual acuity reduced (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3) | 9 (10) | 0 (0) | 2 (2) | 0 (0) | 19 (24) | 35 (41)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 12 (12) | 16 (16)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 6 (7)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Trial Agreement

DOCUMENTS (2):
  • Study Protocol (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/14/NCT02903914/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-21): https://cdn.clinicaltrials.gov/large-docs/14/NCT02903914/SAP_001.pdf